CLINICAL TRIAL: NCT06819540
Title: The Effect of Mindfulness-Based Stress Reduction Programme on Smartphone Addiction, Stress and Quality of Life in University Students
Acronym: Mindfulness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Leyla SEZGİN, Lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 27.12.2024-175288
Record Dates: First submitted 2025-01-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Smartphone Addiction; Mindfulness Based Stress Reduction; Quality of Life
Keywords: Mindfulness; University Students; Stress
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): University students over 18 years of age with smartphone addiction
- experiment (Experimental): University students over 18 years of age with smartphone addiction
  Interventions: Behavioral: Mindfulness-Based Stress Reduction Programme

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction Programme — Mindfulness involves paying attention to what is occurring in the present moment, noticing the particularity of that attention, and accepting without judgement all states of awareness. Mindfulness is important in moving individuals away from automatic thoughts, habits and unhealthy patterns of behaviour, and therefore can play an important role in promoting conscious and self-affirmed behavioural regulation, which has long been associated with enhancing well-being. Mindfulness is a way of regulating one's self, thoughts and awareness. It has been demonstrated to enhance the ability to remain present in the moment, arising through purposeful, momentary, non-judgemental attention to experience. Recently mindfulness appears to have a positive impact on helping people overcome addiction and psychological problems and providing effective techniques to manage them
  Arms: experiment

SUMMARY:
The aim of this observational study was to examine the effect of Mindfulness-Based Stress Reduction Program on Smartphone Addiction, Stress and Quality of Life in Nursing Students. The main question it aims to answer is:

Is there a significant relationship between smartphone addiction, quality of life and stress in nursing students? Smartphone addiction scale will be applied and students with risky scores will be determined and pre-test will be applied to the students in the experimental group according to randomization. During an 8-week intervention period, in addition to mindfulness practices and experiential studies, experiential practices will be carried out on stress, stress management and how mindfulness is applied in daily life and interpersonal communication through the sharing of the participants.

DETAILED DESCRIPTION:
This study was conducted to investigate mindfulness-based stress reduction in nursing students.

To determine the effect of the program on smartphone addiction, stress and quality of life will be carried out for this purpose. The data obtained in the study will only be used in this study. This You will not be charged for the study and you will not receive any remuneration.

Information about you will be kept confidential, but officials overseeing the quality of the study, ethics will be examined if deemed necessary by committees or authorities. Smartphone addiction scale was administered, students with risky scores were identified, and the students who received risky scores were identified during an 8-week intervention period.

in addition to mindfulness practices and experiential work Through the participants' sharing, stress, stress management and mindfulness in daily life and how it is applied in interpersonal communication will be done. After this process is over, the post-test will be applied and necessary analyzes will be made. Education a follow-up test will be performed 12 weeks after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years of age,
* From the highest on the smartphone addiction scale students from the beginning until the sample size is reached
* No diagnosed psychiatric illness or medication not to use it,
* Volunteering to participate in the study
* Muş Alparslan University at the time of the research Continuing education in the Department of Nursing

Exclusion Criteria:

* Students who did not participate in at least two group programs and

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-22 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
6 months improvement in smartphone addiction | 6 months
  Smartphone addiction scale Smartphone Addiction Scale consists of 33 questions. Participants are asked to choose the appropriate option from 'Strongly disagree', 'Disagree', 'Partially disagree', 'Partially agree', 'Agree', 'Strongly agree'. The answers are evaluated between 1-6. The lowest answer score is 33 and the highest answer score is 198. High scorers are those who are seen as risky smartphone users and show addiction. For those with low scores, risky smartphone use is not seen.

SECONDARY OUTCOMES:
6 months improvement in smartphone addiction, stress and quality of life | 6 months
  Perceived Stress Scale (PSS) It consists of 14 items and 2 sub-dimensions. The scale consists of two sub-dimensions: perception of inadequate self-efficacy (4,5,6,7,9,10,13) and perception of stress/discomfort (1,2,3,8,11,12,14). The scale is a five-point Likert-type scale and is evaluated between 'Never: 0', 'Almost Never: 1', 'Sometimes: 2', 'Quite Often: 3', 'Very often (4)'.
  SF-12 Quality of life scale The SF-12, which was transformed into a shorter form by taking 12 different items from 8 different subheadings of the SF-36, consists of two different dimensions: Physical Components Summary Score (PCSS) and Mental Components Summary Score (MCSS). The T-score used to calculate the scoring in SF-36 is not used in SF-12. Instead, a different scoring rule is used. Physical standardisation values and mental standardisation values are summed separately for the answers given by the individuals. Finally, 56.57706 is added to the sum of physical standardisation for 12 questions to calcula